CLINICAL TRIAL: NCT06603636
Title: Foot Progression Angle in Relation to Spatiotemporal Parameters of Gait in Children with Cerebral Palsy
Acronym: FPA
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hisham Elsawy, Clinical researcher, Cairo University
Other Study IDs: P.T.REC/012/002665
Record Dates: First submitted 2024-09-07; First posted 2024-09-19 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Cerebral Palsy (CP)
Keywords: Foot progression angle; Spatiotemporal; Dynamic footprint
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- study group: cerebral palsy children aging from 5 to 8 years having problem in gait

SUMMARY:
The study was applied to assess the difference of the foot progression angle and measuring spatiotemporal parameters of gait among the three age groups (five to six, six to seven and seven to eight years), of diplegic cerebral palsied children and to investigate the relation between FPA of right and left lower extremity and spatiotemporal parameters of gait in diplegic cerebral palsied children.

Sixty diplegic cerebral palsied children from both sexes with age ranged from five to eight years old were participated in this study.

Children were selected from the outpatient clinic of faculty of physical therapy, Cairo University.

They were divided into three equal age groups, group (A) from five to six years, group (B) from six to seven years and group (C) from seven to eight years.

Foot progression angle and spatiotemporal parameters of gait were evaluated for each participated child by the use of dynamic footprint during walking barefoot at free walking speed.

DETAILED DESCRIPTION:
Introduction Cerebral palsy (CP) is the most common pediatric neurological and physical disability. It is a group of permanent disorders of the development of movement and posture that are attributed to non-progressive disturbances that occurred in the developing fetal or infant brain along with accompanying conditions such as mental retardation, epilepsy, perceptual impairment, language impairment, and mental behavior abnormalities.

Foot progression angle (FPA) is defined as the angle between the longitudinal axis of the foot and the line of progression of the child's gait . It represents the rotational gait deviation of the lower extremity from the tip of the femoral head to the foot. It was also defined as the angle of the foot relative to the progressive direction of the subjects during gait .

Abnormal gait is a common problem in children with CP. Because of motor weakness and poor voluntary motor control, crouched gait or diplegic gait is an important functional biomarker in children with spastic diplegic CP. In addition, gait in children with CP is characterized by a slower walking speed, a shorter-stride length, and more time spent in double support .

Purpose of the Study: The purpose of the study is:

To determine the side differences (right and left sides) on FPA values in diplegic CP children from five to eight years.

To measuring spatiotemporal parameters of gait in diplegic CP children from five to eight years.

To investigate the interrelationship between FPA and spatiotemporal parameters diplegic CP children from five to eight years

Subjects, Instrumentations and Procedures

Subjects:

Sixty diplegic and/or hemiplegic CP children will participate in this study. They will be selected from both sexes. Subjects will be selected from the outpatient clinic of Faculty of Physical Therapy, Cairo University according to the following criteria.

Inclusion criteria:

* Their age will be ranged from six to eight years.
* Children diagnosed as diplegic and/or hemiplegic CP.
* Children who can stand and ambulate without the use of an assistive device (At Level II or III on the Gross Motor Function Classification System).
* Their degree of spasticity will be ranged from 1 to 1+ according to the Modified Ashworth Scale.
* Children who are able to follow instructions and understand commands given to them during the testing procedure.
* Dynamic foot print will be used to assess FPA and spatial parameter of gait (step length and stride length).

Exclusion criteria:

* Children with Convulsions.
* Children with fixed contractures of lower extremities.
* Children with surgical interventions in the lower extremities.
* Children with visual and\or auditory disorders.

Instrumentation (materials):

The main used equipment and tools:

1. Modified Ashworth Scale: will be used to determine the degree of spasticity.
2. Gross Motor Function Classification System: will be used to determine children who can stand and ambulate without the use of an assistive device.
3. Dynamic Footprint: Dynamic footprint will be used to measure FPA and spatial parameters of gait. The materials were used for measurement and analyses of FPA (Losel et al., 1996) were:

   • A walkway of 6 m length, 61 cm width and 5 mm height.

   • Paper of 610 cm by 457 cm (20 ft. ×15 ft.) to be placed on the walkway.
   * Adhesive tape to stabilize the paper on the walkway.
   * One chair at each end of the paper.
   * Tray (1 cm depth) large enough to accommodate both feet.
   * Colored powder paint and talcum powder (100:1).
   * Two wet towels.
   * Towel and wet wipes for cleansing feet placed at far end.
   * Artist fixatives spray to be sprayed over successive footprints in order to prevent smudging of the prints.
   * Adhesive transparent contact plastic to be placed over each individual footprint.
   * Scissor for cutting the adhesive tape used to stabilize the paper.
   * Transparent grid (parallel lines).
   * Fine 0.5 mm water soluble pen (non-permanent marker).
   * Two stainless steel rulers (one 30 cm and the other one meter length).
   * Transparent plastic protractor.

   Procedures of the study:

   • Subjects recruitment: Before recruitment, a talk will be given by the researcher to parents to explain the purposes and methodology of the study. The consent forms will then be given to children& parents. After collecting the consent forms, subjects will be examined by the researcher for the inclusion and exclusion criteria. Each eligible child (according to the consent form and examination) will participate in the study.

   The protocol of the study will be explained to the subjects before conducting the study:
   * Dynamic Footprint Procedure:

     1. For measuring FPA:

        This procedure will be classified into two main phases:

     <!-- -->

     1. Measurement phase:

        - Footprint data will be obtained using 6 m lengths of white paper 45 cm wide, for each trail .

        - The paper will be laid out over an elevated walkway 6 m in length and 5 mm above the floor.

        - All lining paper will be affixed with adhesive tape to prevent any slippage during data collection.

        - A chair will be positioned at either end of the paper.

        - The child will not be distracted by anything in the room which may change the motion pattern.

        - Each child will be standing bare-feet and was allowed to walk over the walkway several times to familiarize himself/herself with the procedure.

        - A wet towel will be placed at the base of the chair at both ends.

        - A tray (1 cm depth) large enough to contain both feet, containing a composite mixture of colored powder paint and talcum powder (100:1), at the base of the chair at the starting end, was used to generate the footprints to be analyzed .
        * Each child will be instructed to place both feet on a wet towel, then, to place them in a tray. Excess powder was gently shaken off.
        * The container will be removed and the child was instructed to rise from the chair and walk at free walking speed to the other end, looking straight ahead and sit down upon reaching the other end, for cleansing feet by wet wipes and towel.
        * Once adequate footprint will be obtained, four successive (mid-gait analysis) footprints will be identified to exclude phases of acceleration and deceleration and will be sprayed with artist's fixative spray in order to prevent smearing of the print, and then left to dry.
        * Once dry, a piece of adhesive transparent contact plastic will be placed over each individual footprint before the 6 m length of paper was rolled up.
        * All trails will be laminated to facilitate repeated measurements.
        * Each child's name will be written in each paper.
     2. Analysis phase:

        - The first few steps of the footprints were generally disregarded because they were initiated from a static position, and were therefore not indicative of the subject's steps during active locomotion.

        - A fine 0.5 mm water-soluble pen was used, which enabled marks to be erased and didn't leave any indentations on the laminated surface.

        - Stainless-steel rulers were used to draw lines, and angles were measured with a transparent plastic protractor enabling measurement increments to 0.5°

        - A transparent grid, a simple rectangle made up of parallel lines, was placed over the footprint.

        - The longitudinal border of the grid was aligned with the apex of the hallux and the medial side of the forefoot. To ensure parallel placement of the grid, the distance between the top and bottom margins of the grid and the border of the paper were measured.

        - The grid was used to draw a line (A) representing the apex of the hallux (Figure 2). A similar line (B) was drawn at the posterior aspect of the heel that was parallel to the line (A) dividing the length of the foot into three equal portions and creating lines (C) and (D) (Shores, 1980).
        * The length of line (C) forefoot reference and (D) rear foot reference was measured using the outer borders of the print, each line was bisected and thus midpoints will be determined.
        * The medial and lateral borders of the entire footprint were defined by constructing two lines:

1. The most medial aspect of the forefoot (disregarding the toes) was marked, as was the most medial aspect of the heel. These points were connected by a line to establish the medial border of the print.

2. The most lateral border of the forefoot (again, disregarding the toes) was marked, as was the most lateral border of the heel. These points were connected to establish a lateral border of the print.

The study was applied to assess the difference of the foot progression angle and measuring spatiotemporal parameters of gait among the three age groups (five to six, six to seven and seven to eight years), of diplegic cerebral palsied children and to investigate the relation between FPA of right and left lower extremity and spatiotemporal parameters of gait in diplegic cerebral palsied children.

Sixty diplegic cerebral palsied children from both sexes with age ranged from five to eight years old were participated in this study.

Children were selected from the outpatient clinic of faculty of physical therapy, Cairo University.

They were divided into three equal age groups, group (A) from five to six years, group (B) from six to seven years and group (C) from seven to eight years.

Foot progression angle and spatiotemporal parameters of gait were evaluated for each participated child by the use of dynamic footprint during walking barefoot at free walking speed.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:

  1. Their age will be ranged from six to eight years.
  2. Children diagnosed as diplegic and/or hemiplegic CP.
  3. Children who can stand and ambulate without the use of an assistive device (At Level II or III on the Gross Motor Function Classification System).
  4. Their degree of spasticity will be ranged from 1 to 1+ according to the Modified Ashworth Scale.
  5. Children who are able to follow instructions and understand commands given to them during the testing procedure.
  6. Dynamic foot print will be used to assess FPA and spatial parameter of gait (step length and stride length).

Exclusion Criteria:

1. Children with Convulsions.
2. Children with fixed contractures of lower extremities.
3. Children with surgical interventions in the lower extremities.
4. Children with visual and\or auditory disorders.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: this study were to determine the side differences (right and left sides) on FPA values in diplegic CP children and to measuring spatiotemporal parameters of gait (step length, stride length, speed, cadence, single leg support) in diplegic CP children from five to eight years and to investigate the relation between foot progression angle of right and left lower extremity and spatiotemporal parameters of gait in diplegic cerebral palsied children.
  The study applied at the out clinic of faculty of physical therapy Cairo university
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
foot progression angle | up to 4 months
  Foot progression angle of both right and left foot

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Giza, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: Yes
research results research variables studied number of participants
Supporting Information: Study Protocol
Time Frame: up to 1 months
Access Criteria: any one